CLINICAL TRIAL: NCT00870376
Title: Studies of Biomarkers in Different Urodynamic Diagnoses of Female Patients With Lower Urinary Tract Symptoms
Status: Withdrawn | Type: Observational
Why Stopped: no budget
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 97109
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2015-07

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: lower urinary tract symptoms; biomarkers; urodynamic studies
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- urodynamic studies
  Interventions: Other: biomarkers

INTERVENTIONS:
Other: biomarkers — To define a biomarker or combination of overactive bladder syndrome

SUMMARY:
Urodynamic study is an objective method to evaluate female patients with lower urinary tract symptoms (LUTS). However, this method includes place a urinary catheter, thus prevents it as a routine method to evaluate and follow up patients with LUTS. Therefore, it is necessary to find a simple and objective method to help in evaluating female patients with LUTS. Several kinds of biomarker had been reported in diagnosing patients with overactive bladder; however, the sensitivity remained poor. The aim of this study is to find a useful biomarker, biomarkers, or combinations, with the aid of urodynamic study, to objectively and precisely in evaluating the female patients with LUTS.

ELIGIBILITY:
Inclusion Criteria:

* All female patients (> 20 years) with Lower urinary tract syndrome.

Exclusion Criteria:

* Female patients with tumor and stone were excluded.

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female patients with LUTS
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2009-04-23 (Actual)

PRIMARY OUTCOMES:
The aim of this study is to find a useful biomarker, biomarkers, or combinations, with the aid of urodynamic study, to objectively and precisely in evaluating the female patients with LUTS. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banciao, Taipei, Taiwan